CLINICAL TRIAL: NCT01963299
Title: Prospective Randomised Double-blind Study to Compare Ropivacaine 10mg/mL Alone Versus Ropivacaine 10mg/mL Associated With Clonidine 1µg/kg for Peribulbar Anesthesia in Posterior Eye Surgery
Brief Title: Clonidine - Ropivacaine in Peribulbar Anesthesia
Acronym: CRAPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GIRARD-BERTRAND 2013
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Indication for Surgery of the Posterior Segment Under Locoregional Anaesthesia
MeSH Terms: interventions — Ropivacaine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine alone group (Active Comparator)
  Interventions: Drug: 5 ml Ropivacaine 10% + physiological saline
- Ropivacaine/Clonidine group (Experimental)
  Interventions: Drug: 5 ml Ropivacaine 10% + Clonidine 1 µg/kg

INTERVENTIONS:
Drug: 5 ml Ropivacaine 10% + physiological saline
  Arms: Ropivacaine alone group
Drug: 5 ml Ropivacaine 10% + Clonidine 1 µg/kg
  Arms: Ropivacaine/Clonidine group

SUMMARY:
This is a study conducted in 60 patients, randomly assigned to one of two groups of 30: the first will receive ropivacaine alone and the second will receive the association ropivacaine/clonidine.

The aim of the study is to prove that the association of Clonidine with Ropivacaine is more effective than ropivacaine alone for locoregional anaesthesia of the eye for retinal surgery.

The principal interest of this association of drugs is that it procures faster and longer anaesthesia of the eye with less ropivacaine (therefore fewer injections). This provides greater comfort to the patient during and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients who have given written informed consent
* any adult patient about to undergo their first operation involving the posterior segment of the eye under peribulbar anaesthesia

Exclusion Criteria:

* persons without National Health Insurance
* pregnant or breast-feeding women, patients < 18, patients who cannot give their consent, patient's refusal of Loco-Regional Anesthesia, patients who cannot remain in dorsal decubitus dorsal for at least 1h
* contra-indication for Loco-Regional Anesthesia
* hypersensitivity to the study drugs (ropivacaine, clonidine), to the corresponding excipients or hypersensitivity to local anaesthetics other than amide-type ropivacaine.
* disorders of periorbital or oculomotor sensitivity, patients with glaucoma, patients with chronic pain and on morphines
* uncontrolled arterial hypertension, clonidine per os at home, arterial hypotension before the intervention (SAP < 90 mmHg)
* Surgery for diabetic retinopathy, patients with unbalanced diabetes, eye with prior posterior segment surgery
* Contra-indications mentioned on the summary of product characteristics for clonidine (known hypersensitivity to the active ingredients or one of its excipients, Heart rate below 60bpm, severe Bradycardia due to sinoatrial node disease or second or third degree atrioventricular block, Depression, Sultopride).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08-16 (Actual); Primary Completion 2013-10-07 (Actual); Study Completion 2013-10-07 (Actual)

PRIMARY OUTCOMES:
Dose of ropivacaine injected 10 mg/ml: necessary to obtain complete ocular akinesia | up to 1 hour

SECONDARY OUTCOMES:
Time to achieve akinesia | up to 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France